CLINICAL TRIAL: NCT01903473
Title: Donor Regulatory T Cells (Treg) Infusion (DTI) in Patients With Steroid-refractory Chronic Graft-versus-host Disease (GVHD)
Brief Title: Donor Regulatory T Cells Infusion in Patients With Chronic Graft-versus-host Disease (GVHD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Frédéric Baron, MD, PhD, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TJB1117
Record Dates: First submitted 2013-07-10; First posted 2013-07-19 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Chronic Graft-Versus-Host Disease; Acute Graft-Versus-Host Disease; Steroid Refractory Graft-Versus-Host Disease
Keywords: Allogeneic hematopoietic cell transplantation; GVHD; Regulatory T cells; Steroid refractory; Rapamycin; Immune recovery; Infusion; HLA-identical sibling; HLA-matched unrelated donor; IL-2
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: DTI arm
  * 10 patients will be included in the DTI (Treg) + IL-2 arm.
  * Treg infusion + rapa+ IL-2 will be considered safe if no patients die because of Treg infusion, less than 4 patients die of nonrelapse causes the first 90 days after inclusion in the study, and less than 4 patients experience chronic GVHD progression within the first 90 days after inclusion.
  * The study will be closed at any time a fourth patient experience nonrelapse mortality within 90 days of inclusion or experience GVHD progression within 90 days of inclusion.
  Control arm
  * Up to 25 patients will be included in the control arm.
  * Rapa administration will be considered safe if less than 4/10, 8/20 or 10/25 patients die of nonrelapse causes the first 90 days after inclusion in the study and less than 4/10, 8/20 or 10/25 patients experienced chronic GVHD progression within the first 90 days after inclusion.
  * This arm of the study will be closed at any time the above criteria can no longer be met.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Donor Treg infusion arm (Experimental): Condition:Patients treated with steroids for a chronic GVHD occurring after allogeneic cell transplantation. Patients who have refractory chronic GVHD will be eligible. Patients in this arm will be first treated with Rapamycin while CNI (if any) will be discontinued and infused whith Treg cells 60-90 days after.
  Interventions: Other: T regulatory cells
- Control (Active Comparator): Condition:Patients treated with steroids for a chronic GVHD occurring after allogeneic cell transplantation. Patients who have refractory chronic GVHD will be eligible. Patients in this arm will be treated with Rapamycin which is an alternative immunosupression strategy allowing to fight againt GVHD and CNI (if any) will be discontinued.
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — Rapamycin will be started within 2 weeks after inclusion. Rapamycin will be given at 2-6 mg loading dose for one day, followed by approximately 1 mg daily to achieve a target trough level of 5 to 10 ng/mL. The frequency of trough level measurements will be done according to the investigator choice; Rapamycin may be discontinued in case of resolution of chronic GVHD ≥ 3 months or in case of un-manageable side effects or progression of chronic GVHD.
  Calcineurin inhibitor discontinuation within 2 weeks after rapamycin initiation. No other modification of immunosuppressive drugs and in particular no decrease in the dose of steroids (unless necessary for side effects).
  Other Names: Sirolimus
  Arms: Control
Other: T regulatory cells — One infusion of ≥ 0.5 x10E6 T reg cells/kg recipient at 60-90 days after first day of rapamycin administration and after calcineurin inhibitor discontinuation. The infusion procedure will take one hour.
  Low-dose Il-2 (1x106 IU/day) will be started the day of DTI and will be continued for a period of 2months in order to expand infused donor Tregs.
  Other Names: T suppressor cells; Treg cells
  Arms: Donor Treg infusion arm

SUMMARY:
The immune system has offensive and defensive capacities. In bone marrow transplantation, offensive cells in the donor grafts may attack host's organs, leading to a complication known as Graft versus Host Disease (GVDH). At present, patients receive steroid treatment to combat this tricky situation. Nevertheless, some patients do not respond to this therapy. Recently, it has been shown that immune system cells having defensive capacities can help in preventing the occurrence of a GVDH.

This study aims to evaluate if these protective cells together with a non-standard immunosuppressor can improve the clinical condition and suppress the activity of the offensive cells in the graft.

DETAILED DESCRIPTION:
TREATMENT PLAN

1 Immunosuppressive drugs (DTI and control arms)

* Rapa will be started within 2 weeks after inclusion. Rapa will be given at 2-6 mg loading dose for one day, followed by approximately 1mg daily to achieve a target trough level of 5 to 10 ng/mL. The frequency of trough level measurements will be done according to the investigator choice;
* Rapa may be discontinued in case of resolution of chronic GVHD ≥ 3 months or in case of un-manageable side effects or progression of chronic GVHD.
* Calcineurin inhibitor discontinuation within 2 weeks after rapa initiation. No other modification of immunosuppressive drugs and in particular no decrease in the dose of steroids (unless necessary for side effects).
* Evaluation of chronic GVHD 60 days after rapa initiation. DTI will not be given in patients who had progression of their GVHD on day 60 nor in those who are in CR of their GVHD.

  2. Collection of donor lymphocytes (DTI arm)
* Apheresis of the donor will be performed 60-90 days after first day of rapa administration to the patient.There will be no particular preparation of the donor prior to leukapheresis. After written informed consent, the donor will undergo leukaphereses on 1 day. Leukapheresis will be performed using a continuous flow blood cell separator and following a mononuclear cell collection protocol. The volume of blood processed will be 20 liters. Anticoagulation will be performed with the ACD-A / heparin solution.

  3. Tregselection and infusion (DTI arm)
* Treg will be isolated at the LTCG of the CHU of Liège from apheresis product with the CliniMACS separation system (MiltenyiBiotec) following a two-step procedure (CD8 and CD19 depletion followed by CD25 positive selection)according to the manufacturer's recommendation. Aliquots (≈ 3 mL) of the Treg product will be saved for analyses.
* Treg will be infused i.v.60-90 days after first day of rapa administration and after calcineurin inhibitor discontinuation. No DTI will be performed in the control arm.
* Low-dose Il-2 (1x106 IU/day) will be started the day of DTI and will be continued for a period of 2months in order to expand infused donor Tregs.

PATIENTS' FOLLOW-UP

1. Quality controls of cell products 1.1 Peripheral blood.

   The following laboratory analyses will be performed in the peripheral blood of the donor on the days of lymphocyte collections :
   * Nucleated cell count and differential in an automated cell counter;

   1.1.2 Leukapheresis product as well as start, intermediate, and final fractions of Treg selection.

   The following laboratory analyses will be performed in the lymphocyte collection as well as start, intermediate and final fractions of the Treg selection:

   • Nucleated cell count and differential on an automated cell counter;
   * FACS analysis with determination of the % cells (on total WBC) with the markers: CD20-FITC (Miltenyi #130-091-110), CD14-PE (Miltenyi #130-091-412), CD15-PE (Miltenyi #130-091-390), CD56-PE (Miltenyi #130-090-910), CD45-VioBlue (Miltenyi #130-092-497), CD8-APC (Miltenyi #130-091-083), PropidiumIodid(Miltenyi #130-093-233), T reg Detection Kit (CD4/Cd25/CD127) (Miltenyi #130-096-076), and Treg Detection Kit#2 (CD4/CD25/Foxp3)-APC (Miltenyi #130-094-158).
   * Treg phenotype using the following markers: CD127, CD45RA, CCR4, CCR7 and KI67.
   * Estimation of Treg function42.
   * Methylation status of CpG dinucleotides located in a conserved region of FoxP3 intron
   * Cell viability by trypan blue exclusion.
   * Microbiology testing including standard virology and bacterial culture.

   1.1.3Release criteria.

   The following criteria should be met for release:

   • ≥ 0.5 x106 cells/kg recipient;
   * ≥ 55% CD4+FoxP3+;
   * Viability > 80%;
   * <0.05 x 106 CD45+CD8+ cells/kg.
2. Toxicities of cell infusions Potential toxicities associated with Treg infusions will be carefully monitored per standard procedures.
3. Clinical data

   Patient will be carefully observed and the following clinical parameters will be recorded:

   • Incidence, timing and severity of acute GVHD following DTI, its treatment and outcome;
   * Evolution of chronic GVHD, its treatment and outcome. More specifically, chronic GVHD (including current immunosuppressive therapy) will be assessed for each organ according to the revised NIH consensus:
   * Incidence, timing and severity of secondary cytopenia, its treatment and outcome;
   * Incidence, timing and severity of bacterial, viral, fungal and protozoal infections
   * Duration of hospitalization if any;
   * Evolution of the primary malignant disease: response if not in CR at the time of inclusion, relapse, its treatment and outcome;
   * Any other serious complication associated with the transplant procedure;
   * Death and survival.
4. Immunological data(performed in the GIGA at the ULG for all but the analyses of methylation status of CpG dinucleotides located in a conserved region of FoxP3 intron 1 that will be performed at the UCL).

1) Immune recovery I (flow cytometry). The following analyses will be performed (starting with 5 mL of blood).

2) Immune recovery II. Isolation of T-cell subsets for analyses of repertoire diversity through next-generation sequencing (NGS; starting from 50 mL of blood). The following subsets will be isolated (~50,000 cells each) and then cryopreserved:

* CD4+ CD25+ regulatory T cells (naïve, activated and memory),
* CD4+ CD25- non-regulatory T cells (naïve/memory), and
* CD8+ cytotoxic T cells (naïve/memory).

ELIGIBILITY:
1. Patient criteria : Donor Treg infusion (DTI) and control arms.

* Signed informed consent.
* Grafts from HLA-identical siblings or HLA-matched unrelated donor (1 of 10 HLA-mismatch is allowed).
* ≥ 18 years of age.
* Steroid-refractory or steroid-resistant chronic GVHD defined as:

  * development of 1 or more new sites of disease while being treated for chronic GVHD,
  * progression of existing sites of disease while receiving treatment for chronic GVHD,
  * failure to improve despite at least 1 month of standard treatment for chronic GVHD.

or severe chronic GVHD and contra-indication to the use of steroids and at least failed one prior line of treatment.

* Severe chronic GVHD according to NIH definition.
* No prior failure of rapamycine as treatment for chronic GVHD
* No contra-indication to the use of rapamycin.
* No alemtuzumab administration in the last 6 months.
* GFR > 25 mL/min.
* No HIV seropositivity.
* No fungal infection with radiological progression after treatment with amphotericine B or active azoles for > 1 month.
* No other uncontrolled infection.
* No progression of the hematological malignancy.
* Karnofsky performance score ≥ 70%.
* DLCO > 35% and no need of supplemental continuous oxygen.
* No active post-transplant microangiopathy and no previous microangiopathy while on rapamycine.
* No uncontrolled hypertriglyceridemia.

  2 Donor criteria : DTI arm only.
* Donor ≥ 18 years of age.
* Written informed consent to perform apheresis from the donor (all patients) and permission from the third party donor registry (in case of unrelated donor).
* Standard criteria for leukapheresis and DLI following complete work-up according to standard procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety of a combination of rapa administration, donor Treg infusion and low-dose IL-2 in patients with steroid-refractory chronic GVHD. | 12 months after inclusion
  To assess the immunological changes (including Treg number/phenotype) occurring after donor Treg infusion and rapamycin administration. Treg will be defined as CD4+CD25+FoxP3+ T cells. Treg phenotype will include CD127, CD45RA, CCR4, CCR7 and KI67. Treg will also be assessed by an analysis of the methylation status of CpG dinucleotides located in a conserved region of FoxP3 intron 1.

SECONDARY OUTCOMES:
To assess the efficiency of Treg selection with the Clinimacs procedure. | 1 month after Treg selection
  Treg selection will be performed with the CliniMACS Miltenyi Biotec separation system using a two-step procedure: first, a CD8 and CD19 depletion, followed by CD25 positive selection.
To assess the response rate of chronic GVHD (defined using the NIH criteria as defined by Lee et al.41) to donor Treg infusion + low-dose IL-2 + rapa at 1, 2, 3, 6 and 12 months after rapa onset. | at 1, 2, 3, 6 and 12 months after rapamycin onset
  Using the NIH critera, the response rate of chronic GVHD will be evaluated.
To compare response rate of chronic GVHD in patients given Treg infusion + low-dose IL-2 + rapa (DTI arm) versus in those given rapa without Treg infusion (control arm; vide infra). | at 1, 2, 3, 6 and 12 months after rapamycin onset
  Using the NIH critera, the response rate of chronic GVHD will be evaluated.
To compare the incidence of viral, bacterial, fungal and parasital infection in patients given Treg infusion + low-dose IL-2 + rapa (DTI arm) versus in those given rapa without Treg infusion (control arm; vide infra). | over the 12 months of the trial
  Microbiology testing including standard virology and bacterial culture. In addition fungal and protozoal infections will be sought.
To compare overall relapse incidence in patients given Treg infusion + low-dose IL-2 + rapa (DTI arm) versus in those given rapa without Treg infusion (control arm; vide infra). | 1 year after rapamycin onset
To compare overall survival incidence in patients given Treg infusion + low-dose IL-2 + rapa (DTI arm) versus in those given rapa without Treg infusion (control arm; vide infra). | 1 year after rapamycin onset
To compare overall progression-free survival incidence in patients given Treg infusion + low-dose IL-2 + rapa (DTI arm) versus in those given rapa without Treg infusion (control arm; vide infra). | 1 year after rapamycin onset
To assess the impact of 8 weeks rapamycin administration on percentage and absolute counts of Treg and conventional T cells. | 8 weeks after rapamycin onset
  Specific markers will allow to quantify Treg and conventional T cells
To compare immunological changes in patients given Treg infusion + low-dose IL-2 + rapa (DTI arm) versus in those given rapa without Treg infusion (control arm; vide infra). | Before DTI (day 21-28 after rapamycin onset). Week 1 and 3 after DTI (4-5 anf 6-7 weeks after rapamycin onset); month 3, 6 and 12 after rapamycin onset.
  The comparison will be performed on several sub-populations of CD4+ and CD8+ T cells as well as on various subset of B cells. In addition CMV-specific T cells will be compared between the two treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Baron, MD, PhD, Principal Investigator — CHU-ULg
Locations (2):
- Belgium (2):
  - Katholieke Universiteit Leuven, Leuven, Vlaams-Brabant
  - University Hospital Liège, Liège